CLINICAL TRIAL: NCT01261832
Title: Randomized, Prospective , Open Label, Phase 4 Trial of Efficacy and Safety of Adjunctive Cilostazol in Acute Myocardial Infarction Patients Undergoing Percutaneous Coronary Intervention With Drug-eluting Stent
Brief Title: Efficacy and Safety of Adjunctive Cilostazol in Acute Myocardial Infarction Patients
Acronym: SILOAM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Seung Woon Rha, Associate professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KoreaUGuroH SILOAM
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; Percutaneous coronary intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dual antiplatelet therapy for 1 year (Experimental): Dual antiplatelet therapy for 1 year : dual antiplatelet combination therapy with aspirin and clopidogrel for 1 year
  Interventions: Drug: antiplatelet therapy
- Triple antiplatelet therapy for 1 month (Experimental): Triple antiplatelet therapy for 1 month : triple antiplatelet therapy including cilostazol for 1 month and after then, dual antiplatelet therapy for 11 months
  Interventions: Drug: antiplatelet therapy
- Triple antiplatelet therapy for 6 months (Experimental): Triple antiplatelet therapy for 6 months : triple antiplatelet combination therapy including cilostazol for 6 months and after then, dual antiplatelet therapy for 6 months and cilostazol
  Interventions: Drug: antiplatelet therapy

INTERVENTIONS:
Drug: antiplatelet therapy — Dual antiplatelet therapy is defined as combination therapy with aspirin and clopidogrel and triple antiplatelet therapy is defined as combination therapy with aspirin,clopidogrel and cilostazol.
  Other Names: The brand name of clopidogrel is Plavix.; The brand name of cilostazol is Pletaal.

SUMMARY:
Current antiplatelet therapy in acute coronary syndrome have a focus on the dual antiplatelet therapy including aspirin and clopidogrel. However, the patient's drug resistance of aspirin and clopidogrel is the important cause of poor clinical prognosis. Therefore, recently, clinical research about the triple antiplatelet therapy including cilostazol is actively conducted. But, clinical research about triple antiplatelet therapy for acute myocardial infarction is inadequate situation, and the ideal duration of triple antiplatelet therapy has been actively discussed. Therefore, we try to evaluate the clinical outcomes of triple antiplatelet therapy in acute myocardial infarction patients undergoing percutaneous intervention with drug eluting stent compared with dual antiplatelet therapy and investigate ideal duration of triple antiplatelet therapy through this research.

DETAILED DESCRIPTION:
Drug-eluting stents (DES) have drastically changed the landscape of percutaneous coronary intervention (PCI), with significant reductions in the angiographic restenosis rate and need for repeated revascularization. However, several studies showed that DES is associated with a higher incidence of in-stent thrombosis compared with bare metal stents. Therefore, the latest guideline for antiplatelet therapy after PCI with DES suggests that the dual antiplatelet therapy (aspirin plus clopidogrel) be administered for at least 12 months.But is it enough for high-risk patients? Some studies showed that as many as 50% of the patients who received PCI did not react positively to aspirin or clopidogrel.Furthermore, there is increased platelet activity in acute coronary syndrome, especially in acute myocardial infarction (AMI). compared with aspirin or clopidogrel.A recent study suggested that cilostazol could ameliorate platelet responsiveness to clopidogrel in patients who underwent primary PCI. Furthermore, some other studies showed that the administration of cilostazol after PCI could significantly lower the incidence of in-stent restenosis. Therefore, the present study is designed to evaluate the safety and efficacy of additional administration of cilostazol with aspirin and clopidogrel in a real-world cardiology practice among patients presenting with AMI who received primary PCI with DES.

ELIGIBILITY:
Inclusion Criteria: Acute Myocardial Infarction Undergoing Primary percutaneous coronary intervention.

Exclusion Criteria:

1. The patient has a known hypersensitivity or contraindication to any of the following medications: Heparin, Aspirin, Clopidogrel, Cilostazol
2. Uncontrolled hypertension
3. History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or refuses blood transfusions.
4. Baseline hemogram with Hb<10g/dL or PLT count<100,000/μL
5. Patients already taking warfarin, cilostazol or any other type of anti-platelet agents except aspirin and clopidogrel
6. Gastrointestinal or genitourinary bleeding within the prior 3 months, or major surgery within 2 months.
7. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 951 (Estimated)
Dates: Start 2011-07 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular and Cerebral Events | One Year
  Composite of total death, Nonfatal Myocardial Infarction (Non-QMI , Q-MI), Repeat RevascularizationI (Target Vessel Revascularization +Non Target Vessel Revascularization , Coronary Artery Bypass Graft), Stroke (Ischemic & Hemorrhagic)

SECONDARY OUTCOMES:
Individual outcome of primary end points, Stent thrombosis,Bleeding Complication,PFT (Platelet function test),Genotyping results | One year
  1. Individual outcome of primary end points
  2. Stent thrombosis
  3. Beeding Complication defined by the TIMI criteria & Minor Bleeding, Vascular Complications
  4. Angiographic outcomes at 1 year : Binary restenosis, Late loss, FU MLD, mean % restenosis, restenosis type
  5. IVUS findings at Index and Follow up angiography
  6. PFT (Platelet function test) : at discharge, intercurrent event , after one year
  7. Genotyping results : genetic polymorphism

CONTACTS AND LOCATIONS:
Overall Officials: Seung Woon Rha, MD. PhD., Principal Investigator — Cardiovascular Center, Korea University Guro Hospital, 80, Guro-dong, Guro-gu, Seoul, 152-703, Korea
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

REFERENCES:
- [Background] Chen KY, Rha SW, Li YJ, Poddar KL, Jin Z, Minami Y, Wang L, Kim EJ, Park CG, Seo HS, Oh DJ, Jeong MH, Ahn YK, Hong TJ, Kim YJ, Hur SH, Seong IW, Chae JK, Cho MC, Bae JH, Choi DH, Jang YS, Chae IH, Kim CJ, Yoon JH, Chung WS, Seung KB, Park SJ; Korea Acute Myocardial Infarction Registry Investigators. Triple versus dual antiplatelet therapy in patients with acute ST-segment elevation myocardial infarction undergoing primary percutaneous coronary intervention. Circulation. 2009 Jun 30;119(25):3207-14. doi: 10.1161/CIRCULATIONAHA.108.822791. Epub 2009 Jun 15. PMID 19528339